CLINICAL TRIAL: NCT07251790
Title: PrePAP: Pre-Extubation Continuous Positive Airway Pressure in Very Preterm Infants: A Randomised Controlled Trial
Brief Title: Optimising Breathing Support at Extubation in Very Preterm Infants: A Clinical Study
Acronym: PrePAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Western Health, Australia (Other Government); Royal Women's Hospital, Melbourne, Australia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 120475
Record Dates: First submitted 2025-09-29; First posted 2025-11-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: Infants enrolled in the trial will be randomised to receive one of two extubation procedures, placing them in either the "Extubation with prePAP" arm or the "Extubation without prePAP" arm:
  1. Arm 1: Extubation with prePAP (intervention): nCPAP commenced prior to endotracheal tube removal
  2. Arm 2: Extubation without prePAP (control): nCPAP commenced following endotracheal tube removal
  For both arms, the intervention period will begin with a 2-to-5-minute pre-extubation period (whilst the infant is still ventilated), followed by a post-extubation period of up to 4 hours, and a follow-up period of up to 7 days (168 hours).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extubation with prePAP (Experimental): nCPAP commenced prior to endotracheal tube removal
  Interventions: Procedure: Pre-extubation continuous positive airway pressure
- Extubation without prePAP (No Intervention): nCPAP commenced following endotracheal tube removal

INTERVENTIONS:
Procedure: Pre-extubation continuous positive airway pressure — Prior to extubation (2-to-5 minutes) a CPAP hat will be placed on the infant and the circuit set up. A nasal mask will be applied and nCPAP pressure will be commenced at 10 centimetres of water. Only after nCPAP has been in situ for 2 minutes (maximum 5 minutes) will the endotracheal tube be removed.
  Other Names: PrePAP
  Arms: Extubation with prePAP

SUMMARY:
Many babies born very preterm (<32 weeks of pregnancy) require support to breathe from a breathing machine (mechanical ventilator) via a breathing tube. Although this keeps babies alive, it can damage their lungs. To reduce this damage, doctors and nurses try to change babies to gentler breathing support that does not require a breathing tube. This is usually done using a method called nasal continuous positive airway pressure (nCPAP) that uses a nosepiece to deliver breaths. This process of removing the breathing tube is called "extubation". Many babies will need the breathing tube put back in after extubation (for various reasons) and this is independently associated with poorer outcomes.

This research study aims to compare two ways of performing extubation - both of which are already used regularly by doctors and nurses. The "standard extubation" approach involves taking a baby's breathing tube out first, then applying the nosepiece and starting nCPAP. The more recent approach, called "prePAP", involves applying the nosepiece and starting nCPAP before taking the breathing tube out. Previous research suggests that a prePAP approach may provide better support for babies during extubation. However, larger studies are required before this approach is more commonly used.

This study is investigating whether extubating the baby with prePAP is better than extubating the baby without prePAP.

The main question it aims to answer is: Does initiating nCPAP before extubation in very preterm babies reduce the fall in their oxygen levels post-extubation?

DETAILED DESCRIPTION:
The PrePAP trial will investigate if extubation with prePAP (nCPAP commenced prior to extubation) compared to standard extubation practice (nCPAP commenced after extubation) reduces oxygen desaturation in the four hours immediately post-extubation, in very preterm infants being extubated for the first time within the first 30 days of life.

Many infants born very preterm (<32 weeks' gestation) are intubated at birth to receive respiratory support via invasive ventilation. While essential for survival, invasive ventilation can injure their underdeveloped lungs, disrupt lung development and increase the risk of bronchopulmonary dysplasia, a major cause of long-term respiratory morbidity.

Transitioning infants to non-invasive ventilation as soon as feasible is prioritised by clinicians. However, in very preterm infants, almost 40% of extubation attempts fail due to oxygen desaturation or lung collapse. Re-intubation due to extubation failure can induce further airway injury, cardiovascular instability, and oxygen desaturation, resulting in clinical deterioration and prolonged hospitalisation.

PrePAP has been recently suggested as a method of improving respiratory stability during extubation in preterm infants. PrePAP involves commencing nCPAP prior to extubation, with the intent to maintain lung volumes during extubation; preserving oxygenation from pre- to post-extubation. To date, there isn't any clinical evidence explaining the impact to the lungs when both mechanical ventilation and nCPAP are being applied, nor is there evidence that signals a benefit of using prePAP during extubation. Despite this, prePAP is already used in clinical practice and is described in certain neonatal intensive care unit (NICU) extubation guidelines in Australia.

The PrePAP trial is a prospective, multicentre, unblinded, randomised, controlled trial comparing extubation from mechanical ventilation to nCPAP with and without the application of prePAP in very preterm infants born <30 weeks gestational age at first extubation.

Very preterm infants who meet all inclusion (and no exclusion) criteria will be randomised to receive one of two extubation procedures, placing them in either the "Extubation with prePAP" arm or the "Extubation without prePAP" arm:

1. Arm 1: Extubation with prePAP (intervention): nCPAP commenced prior to endotracheal tube removal
2. Arm 2: Extubation without prePAP (control): nCPAP commenced following endotracheal tube removal

For both arms, the intervention period will begin with a 2-to-5-minute pre-extubation period (whilst the infant is still ventilated), followed by a post-extubation period of up to 4 hours, and a follow-up period of up to 7 days (168 hours). The primary outcome (lowest S/F ratio) is assessed only during the (up to) 4-hour post-extubation period.

The results of this trial will determine the appropriate clinical outcomes and end point for a definitive, larger randomised trial to inform clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The infant is admitted to participating NICU
* The infant is born between 22+0 to 29+6 weeks gestational age
* The infant has been on a form of invasive mechanical ventilation for at least 4 hours
* The infant is being electively extubated for the first time from invasive mechanical ventilation to nCPAP
* The infant is being electively extubated for the first time within 30 days from birth
* The infant is clinically stable (as per clinical and research team consensus)
* The parent(s) or legal guardian(s) provides prospective informed consent.

Exclusion Criteria:

* The infant is born <22 weeks or >30 weeks gestational age
* The infant has a major congenital anomaly involving the cardiac, respiratory or gastrointestinal systems, or a known genetic syndrome or diagnosis that might affect respiratory course and outcomes
* The infant has severe pulmonary hypoplasia due to anhydramnios or oligohydramnios before 22 weeks in which the neonatal clinician anticipates that pulmonary hypoplasia related respiratory failure will be the major respiratory problem in early postnatal life
* The infant is receiving invasive mechanical ventilation via nasotracheal intubation
* The infant is planned for extubation to any other mode of non-invasive respiratory support than nCPAP, or no respiratory support
* Refusal of informed consent from the parent(s), or the infant does not have a guardian who can provide informed consent.

Ages: 0 Hours to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in peripheral oxygen saturation to fraction of inspired oxygen ratio (SF ratio) measured within 4 hours post-extubation, or until escalation to nasal intermittent positive pressure ventilation or re-intubation. | 0 minutes then each minute up to 15 minutes, then every 15 minutes up to 4 hours post-extubation.

SECONDARY OUTCOMES:
CPAP level set at extubation (0 minutes). | Measured during the extubation procedure.
Minimum CPAP level set post-extubation (0 minutes to 4 hours). | Measured from extubation up to 4 hours post-extubation.
Maximum CPAP level set post-extubation (0 minutes to 4 hours). | Measured from extubation up to 4 hours post-extubation.
Incidence of increase in CPAP level post-extubation (0 minutes to 4 hours). | Completed for each participant at 4 hours post-extubation.
Change in peripheral oxygen saturation to fraction of inspired oxygen ratio (SF ratio) measured pre-extubation and within 4 hours post-extubation (-5 minutes to 4 hours). | Measured from 5 minutes pre-extubation up to 4 hours post-extubation.
Change in peripheral oxygen saturation (SpO2) measured pre-extubation and within 4 hours post-extubation (-5 minutes to 4 hours). | Measured from 5 minutes pre-extubation up to 4 hours post-extubation.
Change in fraction of inspired oxygen (FiO2) measured pre-extubation and within 4 hours post-extubation (-5 minutes to 4 hours). | Measured from 5 minutes pre-extubation up to 4 hours post-extubation.
Maximum fraction of inspired oxygen (FiO2) measured pre-extubation and within 4 hours post-extubation (-5 minutes to 4 hours). | Measured from 5 minutes pre-extubation up to 4 hours post-extubation.
Change in incidence of significant oxygen desaturation measured post-extubation (0 minutes to 4 hours). | Measured from extubation up to 4 hours post-extubation.
  Significant oxygen desaturation is defined as SpO2 <80% for >30 seconds
Incidence of escalation to nasal intermittent positive pressure ventilation within 7 days post-extubation. | Completed for each participant at the end of their study period: 7 days post-extubation.
Incidence of re-intubation within 7 days post-extubation. | Completed for each participant at the end of their study period: 7 days post-extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia S Stephen, BBmedSc BBiomedSc(Hons), Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Australia (2):
  - The Royal Women's Hospital, Melbourne, Victoria
  - Joan Kirner Women's and Children's Hospital, Saint Albans, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the PrePAP trial will be available six months after publication of the primary outcome, if the below access criteria are met.
  The study protocol, statistical analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute (MCRI) by emailing georgia.stephen@mcri.edu.au, david.tingay@rch.org.au and mctc@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome.
Access Criteria: Prior to releasing any data the following are required:
  1. A Data Transfer Agreement must be signed between relevant parties.
  2. The MCRI Sponsorship Committee must review and approve your protocol and statistical analysis plan which must include and describe how the data will be used and analysed.
  3. An Authorship Agreement to be agreed to and signed between relevant parties. The Agreement must include details regarding appropriate recognition. Authorship may not be justifiable but some form of acknowledgement is requested.
  4. Agreement to cover any additional costs relating to the provision of the data.
  5. Evidence of ethics approval or waiver of approval, to be compliant with the data transfer agreement and ethics requirements at our end.
  Data will only be shared with a recognised research institution where the MCRI Sponsorship Committee has approved the proposed analysis plan.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Background] Gaertner VD, Ruegger CM. Optimising success of neonatal extubation: Respiratory support. Semin Fetal Neonatal Med. 2023 Oct;28(5):101491. doi: 10.1016/j.siny.2023.101491. Epub 2023 Nov 18. PMID 37993322
- [Background] Bhatia R, Carlisle HR, Armstrong RK, Kamlin COF, Davis PG, Tingay DG. Extubation generates lung volume inhomogeneity in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2022 Jan;107(1):82-86. doi: 10.1136/archdischild-2021-321788. Epub 2021 Jun 23. PMID 34162692
- [Background] Plastina L, Gaertner VD, Waldmann AD, Thomann J, Bassler D, Ruegger CM. The DELUX study: development of lung volumes during extubation of preterm infants. Pediatr Res. 2022 Jul;92(1):242-248. doi: 10.1038/s41390-021-01699-w. Epub 2021 Aug 31. PMID 34465873